CLINICAL TRIAL: NCT04240756
Title: 2/2 Treating Mothers with ADHD and Their Young Children Via Telehealth: a Hybrid Type I Effectiveness-Implementation Trial
Brief Title: Treating Parents with ADHD and Their Young Children Via Telehealth: a Hybrid Type I Effectiveness-Implementation Trial
Acronym: TPAC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: Children's National Research Institute (Other); University of Michigan (Other); Seattle Children's Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrea Chronis-Tuscano, Professor, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01MH118320 (NIH); 1R01MH118313 (NIH)
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: ADHD; Parenting
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parent Stimulant Medication + Child Treatment Strategy (Experimental): Parent stimulant medication first followed by a child treatment strategy consisting of behavioral parent training followed by a recommendation for child stimulant medication to the primary care provider if the child remains impaired.
  Interventions: Behavioral: Behavioral Parent Training; Drug: Extended release mixed amphetamine salts (MAS)
- Child Treatment Strategy (Active Comparator): Child treatment strategy consisting of behavioral parent training followed by a recommendation for child stimulant medication to the primary care provider if the child remains impaired. In this arm, parents do not receive stimulant medication before behavioral parent training.
  Interventions: Behavioral: Behavioral Parent Training

INTERVENTIONS:
Behavioral: Behavioral Parent Training — Parents will receive 10 sessions of behavioral parent training with components specifically targeted toward parents with ADHD. Treatment will be delivered via telehealth.
Drug: Extended release mixed amphetamine salts (MAS) — The MAS protocol will include a 2-4 -week open-label titration beginning at 20 mg and dose level will be increased weekly at telehealth visits with the psychopharmacologist until an optimal response or maximum dose of 60 mg.
  Arms: Parent Stimulant Medication + Child Treatment Strategy

SUMMARY:
This study will compare the effectiveness of combined parental stimulant medication and behavioral parent training (BPT) versus BPT alone on child ADHD-related impairment (primary outcome), child ADHD and externalizing symptoms, time to child stimulant prescription (secondary child outcomes) and parental ADHD impairment, parental ADHD symptoms, parenting, and BPT engagement (parental outcomes/target mechanisms). This study will also assess the care delivery context and develop an implementation approach for treatment of families with a parent with ADHD and a child with elevated ADHD symptoms via telehealth in primary care sites providing pediatric care.

DETAILED DESCRIPTION:
Parental ADHD, present in 25-50% of families of children with ADHD and frequently untreated, interferes with effective parenting and predicts poor child developmental and behavioral treatment outcomes. Based on the literature and our own pilot data, the study will randomly assign parents with ADHD and their young at-risk children to one of two conditions: (1) stimulant medication for parents with ADHD followed by a child treatment strategy (CTS) beginning with behavioral parent training (BPT) with the added recommendation of child stimulant treatment if the child remains impaired or (2) a CTS without treatment for parental ADHD. The study will compare treatment effects on child ADHD-related impairment (primary outcome), child ADHD and externalizing symptoms, and time to child stimulant prescription (secondary child outcomes). The study will also examine target mechanisms including improvements in parental ADHD-related impairment and symptomatology (attention, impulsivity, emotional regulation), parenting skills, and BPT engagement, as well as treatment moderators (baseline parental ADHD severity, parental impairment, and parenting skills). Moreover, in an effort to develop a model of treatment that has potential for widespread dissemination while also reducing barriers to receiving care, the study will examine an implementation model involving parent ADHD screening in primary care followed by collaborative care delivered by co-located mental health providers via telehealth. Further, the investigators will develop an implementation plan and associated toolkit using a stakeholder participatory strategy to enhance the ability to move efficiently to adoption of this approach. In addition, the investigators will study the care delivery context, assessing procedures for and rates of screening and participation as well as staffing, workflow, provider- and patient-level acceptability, readiness, and feasibility of implementation approaches. This hybrid effectiveness-implementation project will be achieved via a collaborative R01 across 2 research sites in the US (N = 240 families), with 4-5 primary care partners at each site.

ELIGIBILITY:
Child Inclusion Criteria:

* Be at least 3 years old and no more than 8 years old
* ADHD medication naive or have not had an adequate trial of stimulant medications
* Have ≥5 inactivity or ≥5 hyperactivity symptoms rated as 1 or 2 on the Vanderbilt
* Have a CGI-S-ADHD rating ≥4 and <7

Child Exclusion Criteria:

* Severe ADHD (CGI-S-ADHD score of greater than 6)

Parent Inclusion Criteria:

* Be at least 21 years old and English-speaking
* Meet full DSM-5 criteria for ADHD (any subtype)
* Have findings on physical examination, laboratory studies, vital signs, and electrocardiogram judged to be normal for age with no contraindications for stimulant medication
* Have pulse and blood pressure (BP) within 95% of age and gender mean
* Women of childbearing potential agree to use a medically accepted contraception method consistently
* Parents with common comorbid conditions will be included provided that: (a) they do not report active suicidal ideation with intent (i.e. Beck Depression Inventory (BDI)-II score of 2 or 3 to Q9 which assesses suicidal thoughts); and (b) if receiving an antidepressant medication, their medication is well-tolerated, has not changed within 30 days, and the prescribing physician approves of their participation in the study
* Must have regular access to a computer or phone that can be used to deliver the behavioral parent training

Parent Exclusion Criteria:

* History of allergic or other severe negative reactions to study medications
* Substance abuse in the past 3 months, or a positive baseline urinary toxic screen that is not explained by a time-limited medical circumstance
* Current bipolar disorder, schizophrenia, psychoses, or other primary psychiatric disorder requiring other immediate treatment
* History of chronic/acute medical disorder for which stimulant therapy would be contraindicated (e.g., glaucoma, hypertension)
* Stimulant medication for ADHD in the past 30 days
* Is pregnant

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in child ADHD-related impairment | Baseline, 16 weeks, 36 weeks
  Assessed using the Clinical Global Impressions (CGI) - Attention-Deficit/Hyperactivity Disorder (ADHD) - Severity scale. Minimum value = 1, maximum value = 7. Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Chronis-Tuscano, Ph.D., Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The study data will be shared via the National Database for Clinical Trials related to Mental Illness (NDCT) and will be posted on clinicaltrials.gov upon completion of the grant.
Time Frame: The NFCT will be updated every 6 months and all of the data will be added to clinicaltrials.gov upon completion of the grant.

REFERENCES:
- [Background] Chronis-Tuscano A, Seymour KE, Stein MA, Jones HA, Jiles CD, Rooney ME, Conlon CJ, Efron LA, Wagner SA, Pian J, Robb AS. Efficacy of osmotic-release oral system (OROS) methylphenidate for mothers with attention-deficit/hyperactivity disorder (ADHD): preliminary report of effects on ADHD symptoms and parenting. J Clin Psychiatry. 2008 Dec;69(12):1938-47. doi: 10.4088/jcp.v69n1213. Epub 2008 Dec 2. PMID 19192455
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Schoenfelder EN, Chronis-Tuscano A, Strickland J, Almirall D, Stein MA. Piloting a Sequential, Multiple Assignment, Randomized Trial for Mothers with Attention-Deficit/Hyperactivity Disorder and Their At-Risk Young Children. J Child Adolesc Psychopharmacol. 2019 May;29(4):256-267. doi: 10.1089/cap.2018.0136. Epub 2019 Apr 13. PMID 30950637
- [Background] Chronis-Tuscano A, Rooney M, Seymour KE, Lavin HJ, Pian J, Robb A, Efron L, Conlon C, Stein MA. Effects of maternal stimulant medication on observed parenting in mother-child dyads with attention-deficit/hyperactivity disorder. J Clin Child Adolesc Psychol. 2010;39(4):581-7. doi: 10.1080/15374416.2010.486326. PMID 20589568
- [Background] Chronis-Tuscano A, O'Brien KA, Johnston C, Jones HA, Clarke TL, Raggi VL, Rooney ME, Diaz Y, Pian J, Seymour KE. The relation between maternal ADHD symptoms & improvement in child behavior following brief behavioral parent training is mediated by change in negative parenting. J Abnorm Child Psychol. 2011 Oct;39(7):1047-57. doi: 10.1007/s10802-011-9518-2. PMID 21537894
- [Background] Chronis-Tuscano A, Wang CH, Woods KE, Strickland J, Stein MA. Parent ADHD and Evidence-Based Treatment for Their Children: Review and Directions for Future Research. J Abnorm Child Psychol. 2017 Apr;45(3):501-517. doi: 10.1007/s10802-016-0238-5. PMID 28025755
- [Derived] Lui JHL, Danko CM, Triece T, Bennett IM, Marschall D, Lorenzo NE, Stein MA, Chronis-Tuscano A. Screening for parent and child ADHD in urban pediatric primary care: pilot implementation and stakeholder perspectives. BMC Pediatr. 2023 Jul 13;23(1):354. doi: 10.1186/s12887-023-04082-2. PMID 37442955